CLINICAL TRIAL: NCT01187693
Title: The Outcome Effect of Shoe Lift for Individuals With Low Back Pain and Pronated Foot Due to Anatomical Leg Length Discrepancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Huei-Ming Chai, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 201006053R
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Low Back Pain; Flatfoot; Leg Length Inequality
MeSH Terms: conditions — Low Back Pain; Flatfoot; Leg Length Inequality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shoe lift (Other)
  Interventions: Other: shoe lift

INTERVENTIONS:
Other: shoe lift — shoe lift for balancing the heights of bilateral pelvis of participants with leg length discrepancy during standing

SUMMARY:
People with anatomical leg length discrepancy (LLD) commonly presented excessive subtalar pronation of the long leg compared to their short leg in order to equalize leg length. Although such compensation may decrease the stress in the pelvis and/or low back region, the pronated foot may lead to excessive stress loading onto the ankle or foot, resulting in musculoskeletal injuries. Clinically, the pronated foot has been effectively controlled using functional orthoses with proper posting by adjusting the subtalar joint in the neutral position. But for people with compensatory pronated foot resulted from anatomical LLD, to control excessive pronation of the long leg would exaggerate their asymmetry in leg length. Instead, the pronated foot can be controlled simply by adjusting the length of the short leg. However, there is limited evidence of such intervention in previous literature. The purpose of this research project is going to determine the effect of leg length adjustment on pronation control in people with anatomical LLD. According to this purpose, 5 study objectives will be developed: 1) to examine the validity and reliability of LLD measurement using a hand-held laser distance meter, 2) to compare the foot types before and after leg length adjustment, 3) to compare the kinetic variables before and after leg length adjustment during quiet stance, 4) to compare the kinetic variables before and after leg length adjustment during level walking, and 5) to compare symptoms and functional levels related to low back pain (LBP) before and after leg length adjustment.

The present research project will be designed as a convenience sampling, prospective, quasi-experimental, and pretest/posttest design. There will be 2 parts in this research: 1) validity and reliability test of laser measure for leg length and 2) foot morphology and kinetic analysis before and after leg length adjustment. For the first part of this research, 10 male adults and 20 adults will be recruited for the validity and reliability tests respectively. Anthropometric measurements, including body height, body weight, foot length, foot width, and heel-ball distance, will be measured after a consent form is signed. Participants of the validity test will receive standing pelvic radiography and laser measure to measure their leg length. Each participant of the reliability test will receive 2 sessions of laser measure using a hand-held laser-distance meter. For the first session, all laser measurements will be employed twice by 2 raters with a rest interval of more than 5 min. One week later, another session of laser measure will be given again by one of these 2 raters. Intraclass correlation coefficient (ICC) will be used to test the interrater reliability, intrarater reliability, and validity of the laser measure method. Standard error of measurement (SEM), and small real difference (SRD) will be calculated to represented intrarater reliability also. For the second part of the research, another thirty adults with compensatory pronated foot resulted from LLD will be included in the research project but the sample size will be adjusted to the appropriate number according to power analysis. Each participant will be asked to fill out the visual analog scale (VAS) and the Oswestry Disability Index (ODI) and receive tests containing foot type examination, quiet stance with eye opening, quiet stance with eye closed, and level walking. All tests will be performed before and after leg length adjustment. The experiment will be completed after collecting 3 successful trials for each test. All procedures will be done one month later. ANOVA with repeated measures will be calculated to compare the differences in these variables among before, immediately after, and 1 month following leg length adjustment when the data fit the assumptions of normal distribution. Discrete variables or variables with non-normal distribution were tested using the Friedman test. All statistical analyses will be calculated using SAS 9.1.3. The significant level was set at α = 0.05 while the power was at 0.8.

Five possible results may be expected from conducting this research project: 1) there will be good validity and reliability of the laser distance meter to measure LLD, 2) there will be significant differences in measurements of foot type before and after leg length adjustment, 3) there will be significant differences in kinetic data during quiet stance before and after leg length adjustment, 4) there will be significant differences in kinetic data during level walking before and after leg length adjustment, and 5) symptom and functional level related to LBP will improve after leg length adjustment. Completion of this research project will be projected to provide solid and objective evidences for leg length adjustment through views of morphology and kinetics in people with pronated foot due to anatomical LLD.

ELIGIBILITY:
Inclusion Criteria:

* Leg length discrepancy between 0.5~2 cm
* Chronic low back pain
* Pronated foot of the longer leg (the magnitude of pronation should be more of the longer leg than of the short)

Exclusion Criteria:

* History of operation in low back, pelvis, and lower extremities
* Severe deformity of lower extremities
* Sacroiliac dysfunction
* Symptoms or diseases of neural system
* History of osteoarthritis in lower extremities
* History of sciatica
* History of herniated intervertebral disc
* History of spondylolysis
* History of spondylolisthesis
* History of trauma in the low back
* History of compression fracture in lumbar spine
* History of ankylosing spondylosis
* People have received shoe insole intervention in recent 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
ground reaction force | one month

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Ming Chai, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- School and Graduate Institute of Physical Therapy National Taiwan University, Taipei, Taipei, Taiwan